CLINICAL TRIAL: NCT05088239
Title: Division of Plastic and Reconstruction Surgery
Brief Title: Deep Inferior Epigastric Artery Flap for Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CYCH-IRB No.2020092
Record Dates: First submitted 2021-10-06; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Perforator Flap; Anti-Infectives Adverse Reaction; Infections
Keywords: Prophylatic antibiotics; DIEP flap
MeSH Terms: conditions — Breast Neoplasms; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PAD: In prophylactic antibiotics for drain group (PAD) (n = 15), prophylactic cefazolin 1000 mg was given 30 minutes before surgery, every 4 hours in the peri-operative period, and every 6 hours in the post-operative for 10-14 days when the drains were removed from the breast and abdomen.
  Interventions: Drug: prophylactic antibiotics duration
- PA3: In the 3-day prophylactic antibiotics group (PA3) (n = 11), prophylactic cefazolin 1000 mg was given 30 minutes before surgery, every 4 hours in peri-operative period, and 6-hourly thereafter for 3 days.
  Interventions: Drug: prophylactic antibiotics duration
- PA1: In the 1-day prophylactic antibiotics group (PA1) (n = 82), patients received prophylactic cefazolin 1000 mg 30 minutes before surgery, every 4 hours in the peri-operative period, and every 6 hours in the post-operative period and antibiotics were discontinued within 24 hours of surgery.
  Interventions: Drug: prophylactic antibiotics duration

INTERVENTIONS:
Drug: prophylactic antibiotics duration — Prophylactic cefazolin 1000 mg was given 30 minutes before surgery, every 4 hours in the peri-operative period, and every 6 hours in the post-operative care. Different discontinued duration of antibiotics was divided to 3 groups in one day, 3 days and until to drain removal.

SUMMARY:
Background: There is no consensus on the duration of prophylactic antibiotics for autologous breast reconstruction after mastectomy. We try to standardize prophylactic antibiotics use during breast reconstruction with deep inferior epigastric perforator flap following mastectomy.

Methods: This retrospective case series involved 108 patients who underwent immediate breast reconstruction with deep inferior epigastric perforator flap in Ditmanson Medical Foundation Chia-Yi Christian Hospital between 2012 and 2019. Patients were divided into three groups based on prophylactic antibiotic duration: 1 day, 3 days and >7 days for patients with drains Data were analyzed between January and April, 2021.

ELIGIBILITY:
Inclusion Criteria:

* This retrospective study involved 108 patients who underwent immediate DIEP flap breast reconstruction after unilateral or bilateral mastectomy at the Ditmanson Medical Foundation Chia-Yi Christian Hospital between 2012 and 2019.

Exclusion Criteria:

* Age < 20 years old.

Ages: 24 Years to 63 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This retrospective study involved 108 patients who underwent immediate DIEP flap breast reconstruction after unilateral or bilateral mastectomy at the Ditmanson Medical Foundation Chia-Yi Christian Hospital between 2012 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
surgical site infection (SSI) | Patients were then followed up in the outpatient department for 1 year.
  Infection rate of surgical wounds of breast and abdomen.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Liang Fang, Director, Study Director — Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chia-Yi City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Prophylactic antibiotics discontinued within 24 hours after deep inferior epigastric perforator flap reconstruction can prevent surgical site infection occurrence.